CLINICAL TRIAL: NCT00436098
Title: Pediatric Exercise With Congenital Heart Defects (Kinderturnen Mit Angeborenem Herzfehler)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Collaborators: Lehrstuhl für Präventive und Rehabilitative Sportmedizin der TU Muenchen (Unknown); Kuratorium für Prävention und Rehabilitation an der TU Muenchen (Unknown)
Responsible Party: Dr. A Hager, Deutsches Herzzentrum Munich
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GE IDE No. H00107
Record Dates: First submitted 2007-02-15; First posted 2007-02-16 (Estimated); Last update posted 2008-08-27 (Estimated); Status verified 2008-08

CONDITIONS: Heart Defects, Congenital
Keywords: congenital heart disease; exercise training; motorpedagogical exercise; children; CHD: hemodynamically not significant defects; CHD: acyanotic defects after repair; CHD: cyanotic defects after repair
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): physical training
  Interventions: Behavioral: Motorpedagogic exercise
- 2 (No Intervention)

INTERVENTIONS:
Behavioral: Motorpedagogic exercise — physical training
  Arms: 1

SUMMARY:
Children with congenital heart defects have shown to develop motor coordinative deficiencies. In this study we want to show that a motor pedagogic physical training can improve the coordinative capabilities of children aged 4-6 years.

DETAILED DESCRIPTION:
The study will be performed with a randomized crossover design. After the first assessment of coordinative capabilities children were randomized into two groups. One starts with exercised training for three months. After midterm assessment of the capabilities they will pause for another 3 months and reassessed. The second group will start without training for the first three months. After midterm assessment they will train for three months and have their final assessment.

ELIGIBILITY:
Inclusion Criteria:

* without significant residuals hemodynamically not significant
* without significant residuals after repair
* age 4-6 incl.

Exclusion Criteria:

* gradient at coarctation site > 20 mmHg
* gradient RVOT, PV, LVOT, or AoV > 30 mmHg
* right-left shunt (rest or exercise)
* left-right shunt with dilatation or failure of ana cardiac chamber
* pulmonary hypertension
* heart failure, necessitating therapy
* (suspected) myocarditis or cardiomyopathy
* significant arrhythmia
* ion channel defects, other arrhythmic diseases
* Fontan-like circulation
* repair by atrial switch
* oral anticoagulation
* other medical problems curtailing exercise capacity

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2007-02; Primary Completion 2009-11 (Estimated); Study Completion 2010-05 (Estimated)

PRIMARY OUTCOMES:
Activity: triaxial accelerometry | 3 months

SECONDARY OUTCOMES:
coordinative test: MOT 4-6 | 3 months
coordinative test: LOS KF 18 | 3 months
Quality of life: Kiddy-KINDL | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Alfred Hager, MD, Principal Investigator — Deutsches Herzzentrum München
Locations (2):
- Germany (2):
  - Deutsches Herzzentrum Muenchen, Munich
  - Kuratorium für Prävention und Rehabilitation der TU München, Munich